CLINICAL TRIAL: NCT04438603
Title: The Applicaiton of Immune Repertoire in the Diagnosis and Disease Monitoring of IgA Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: RenJi Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XHEC-C-2020-070-1
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: IgA Nephropathy
Keywords: IgA Nephropathy; IR-Seq; Biomarker
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples; Blood samples taken using PAXgene vacuum blood collection tubes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- IgAN patients at low risk of disease progression: n = 30, incipient disease
  Interventions: Drug: Intervention for incipient patients at low risk of disease progression
- IgAN patients at high risk of disease progression: n = 60, incipient disease
  Interventions: Drug: Intervention for patients at high risk of disease progression
- Long-term stable patients: n = 30, follow-up for at least 15 years
- Progressive IgAN patients: n = 30
- Healthy control: n = 30

INTERVENTIONS:
Drug: Intervention for incipient patients at low risk of disease progression — Conservative treatment, if necessary use ACEI/ARB and titrated to the maximum tolerated dose, with a BP-lowering goal of < 130/80 mm Hg
  Groups: IgAN patients at low risk of disease progression
Drug: Intervention for patients at high risk of disease progression — BP-lowering goal of < 125/75 mm Hg and treat with steroids or steroids combined with immunosuppressants based on optimal supportive therapy:
  1. If GFR>60 ml/min/1.73m^2, oral prednisone 0.6-0.8 mg/kg/day ( (maximum dose 48 mg/day) for 2 months, followed by a monthly dose reduction of 8 mg for 24 weeks.
  2. If GFR is 30-60 ml/min/1.73m^2, intravenous cyclophosphamide (CTX) 750 mg per month per m^2 for 6 months, along with oral prednisone (at the same dose as 1); if intravenous administration is unacceptable, then the above regimen was replaced with oral mycophenolate mofetil 500 mg bid for 24 weeks.
  Groups: IgAN patients at high risk of disease progression

SUMMARY:
This prospective study aims to investigate the role of IR-Seq in the diagnosis and disease monitoring in patients with IgA nephropathy.

DETAILED DESCRIPTION:
Autoimmunity may play an important role in IgA nephropathy, and previous studies have shown that immune repertoire sequencing (IR-Seq) may help elucidate the dynamic changes of immune repertoire (IR) in autoimmune disease states. To further explore the potential application value of this technology, we will conduct a series of prospective studies to investigate the role of IR-Seq in the diagnosis and disease monitoring in patients with IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. IgA nephropathy:

1. Age: 18-80 years.
2. Patients diagnosed with primary IgA nephropathy by renal biopsy.
3. Estimated glomerular filtration rate (using the 2009 CKD-EPI formula) ≥30ml/min/1.73/m^2.
4. Obtain informed consent from patients. 2. Healthy Control: Gender, age and ethnicity matched health volunteers. 3. IgAN patients were further divided into 4 groups, as defined below:

1) Long-term stable patients:

Follow-up for at least 15 years and meet at least one of the following:

1. Annual eGFR loss rate <3ml/min/1.73m^2.
2. eGFR>90ml/min/1.73m^2. 2) Non-progressive IgAN patients:

Meet at least one of the following:

1. eGFR decrease of more than 50% from baseline (in the absence of other possible causes of kidney damage).
2. Annual eGFR loss rate >5ml/min/1.73m^2.
3. Progress to ESRD. 3) IgAN patients at low risk of disease progression: Proteinuria ≤ 1g/24h after 3 months of optimized supportive care. 4) IgAN patients at high risk of disease progression: Proteinuria > 1g/24h despite 3 months of optimized supportive care.

Exclusion Criteria:

1. Kidney biopsy shows crescentic IgAN or MCD-IgAN.;
2. Patients with secondary IgAN;
3. During pregnancy or lactation;
4. After kidney transplantation;
5. More than one serious acute infection in the psat 12 months;
6. Chronic infection;
7. Use of glucocorticosteroids and other immunosuppressive drugs within the last 6 months;
8. Incomplete medical history or clinical data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University Affiliated Sixth People's Hospital, RenJi Hospital, Shanghai Zhongshan Hospital, Longhua Hospital Shanghai University of Traditional Chinese Medicine and Shanghai East Hospital
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Urinary protein remission rate | 24 weeks
  Including complete and partial remission rate of urinary protein. Complete remission criteria: post-treatment urine protein <0.3 g/24h; partial remission criteria: post-treatment urine protein <50% of the maximum value.

SECONDARY OUTCOMES:
24-hour urine protein level | 24 weeks
Serum albumin level | 24 weeks
eGFR (estimated using the 2009 CKD-EPI formula) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China